CLINICAL TRIAL: NCT07361510
Title: ROSETTA Lung-202: A Randomized, Double-Blind, Phase 3 Study of Pumitamig Monotherapy Compared to Pembrolizumab as First-line Treatment in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With PD-L1 ≥ 50%.
Brief Title: A Study to Evaluate the Efficacy of Pumitamig Versus Pembrolizumab in Participants With Previously Untreated Advanced Non-Small Cell Lung Cancer and PD-L1 ≥ 50%. (ROSETTA Lung-202)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA266-0002; 2025-523586-18 (Other: EU CT Number); U1111-1326-9286 (Other: UTN)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Non-Small Cell Lung Cancer (NSCLC); 1L NSCLC; Programmed death ligand-1 (PD-L1); Frst line NSCLC; Advanced NSCLC; Metastatic NSCLC; Pumitamig; Pembrolizumab; ROSETTA LUNG-202; ROSETTA LUNG; CA2660002
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Pumitamig (Experimental)
  Interventions: Drug: Pumitamig
- Arm B: Pembrolizumab (Active Comparator)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pumitamig — Specified dose on specified days
  Other Names: BMS-986545
  Arms: Arm A: Pumitamig
Drug: Pembrolizumab — Specified dose on specified days
  Arms: Arm B: Pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the efficacy of Pumitamig versus Pembrolizumab in participants with previously untreated advanced Non-Small Cell Lung Cancer and PD-L1 ≥ 50%.

ELIGIBILITY:
Inclusion Criteria

* Participants must have a histologically or cytologically confirmed diagnosis of Non-Small Cell Lung Cancer (NSCLC) (squamous and nonsquamous) with Stage IIIB/IIIC or Stage IV disease.
* Participants must have a programmed death ligand-1 (PD-L1) expression ≥ 50%.
* Participants must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Participants must have no prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.

Exclusion Criteria

* Participants must not have any documented actionable genomic alteration (AGA) for which first-line (1L) approved therapies are indicated.
* Participants must not have any symptomatic untreated central nervous system (CNS) metastases, leptomeningeal metastases (carcinomatous meningitis) or spinal cord compression.
* Participants must not have any significant cardiovascular impairment as evidenced by uncontrolled hypertension (despite optimal medical treatment), congestive heart failure, active coronary disease (within 6 months prior to randomization), ventricular arrhythmias, or major thrombotic or embolic events or major hemorrhagic events (within 6 months prior to randomization), or significant risk of pulmonary hemorrhage.
* Participants must not an active autoimmune disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2026-04-09 (Estimated); Primary Completion 2031-10-14 (Estimated); Study Completion 2031-10-14 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) by Blinded Independent Central Review (BICR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 3 years
Overall survival (OS) | Up to approximately 5 years

SECONDARY OUTCOMES:
PFS by investigator according to RECIST v1.1 | Up to approximately 3 years
Objective Response (OR) by BICR according to RECIST v1.1 | Up to approximately 3 years
Duration of response (DOR) by BICR according to RECIST v1.1 | Up to approximately 3 years
Disease control rate (DCR) by BICR according to RECIST v1.1 | Up to approximately 3 years
Time to Response (TTR) by BICR according to RECIST v1.1 | Up to approximately 3 years
Time to definitive deterioration (TTDD) based on the Non-Small Cell Lung Cancer-Symptom Assessment Questionnaire (NSCLC-SAQ) defined as the time from randomization until a definitive clinically meaningful worsening in symptoms or in NSCLC-SAQ total score | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (250):
- United States (32):
  - Local Institution - 0348, Mobile, Alabama
  - Local Institution - 0391, Glendale, Arizona
  - Local Institution - 0352, Beverly Hills, California
  - Local Institution - 0299, Fountain Valley, California
  - Local Institution - 0027, Los Alamitos, California
  - Local Institution - 0208, Pleasant Hill, California
  - Local Institution - 0340, Lakewood, Colorado
  - Local Institution - 0192, Clermont, Florida
  - Local Institution - 0395, Miami, Florida
  - Local Institution - 0355, Palm Bay, Florida
  - Local Institution - 0284, Douglasville, Georgia
  - Local Institution - 0160, Boise, Idaho
  - Local Institution - 0289, Lexington, Kentucky
  - Local Institution - 0350, Columbia, Missouri
  - Local Institution - 0224, Laurelton, New York
  - Local Institution - 0026, New York, New York
  - Local Institution - 0214, Westbury, New York
  - Local Institution - 0300, Pinehurst, North Carolina
  - Local Institution - 0283, Winston-Salem, North Carolina
  - Local Institution - 0383, Cincinnati, Ohio
  - Local Institution - 0288, Lancaster, Pennsylvania
  - Local Institution - 0028, Pittsburgh, Pennsylvania
  - Local Institution - 0344, York, Pennsylvania
  - Local Institution - 0376, Galveston, Texas
  - Local Institution - 0353, Houston, Texas
  - Local Institution - 0351, San Antonio, Texas
  - Local Institution - 0381, San Antonio, Texas
  - Local Institution - 0337, Richmond, Virginia
  - Local Institution - 0349, Winchester, Virginia
  - Local Institution - 0384, Spokane, Washington
  - Local Institution - 0339, Charleston, West Virginia
  - Local Institution - 0380, Green Bay, Wisconsin
- Argentina (5):
  - Local Institution - 0076, Mar del Plata, Buenos Aires
  - Local Institution - 0229, Rosario, Santa Fe Province
  - Local Institution - 0362, Rosario, Santa Fe Province
  - Local Institution - 0058, Buenos Aires
  - Local Institution - 0374, Córdoba
- Australia (6):
  - Local Institution - 0360, Kanwal, New South Wales
  - Local Institution - 0176, Penrith, New South Wales
  - Local Institution - 0154, Elizabeth Vale, South Australia
  - Local Institution - 0221, Ballarat, Victoria
  - Local Institution - 0201, Epping, Victoria
  - Local Institution - 0038, Joondalup, Western Australia
- Austria (3):
  - Local Institution - 0064, Linz, Upper Austria
  - Local Institution - 0196, Feldkirch
  - Local Institution - 0095, Sankt Pölten
- Belgium (4):
  - Local Institution - 0345, Brasschaat, Antwerpen
  - Local Institution - 0333, Auderghem, Bruxelles-Capitale, Région de
  - Local Institution - 0109, Leuven, Vlaams-Brabant
  - Local Institution - 0188, Edegem
- Brazil (7):
  - Local Institution - 0148, Fortaleza, Ceará
  - Local Institution - 0066, Natal/RN, Rio Grande do Norte
  - Local Institution - 0245, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0085, Barretos, São Paulo
  - Local Institution - 0375, São Paulo, São Paulo
  - Local Institution - 0090, Taubaté, São Paulo
  - Local Institution - 0163, São Paulo
- Bulgaria (4):
  - Local Institution - 0202, Rousse
  - Local Institution - 0326, Sofia
  - Local Institution - 0047, Sofia
  - Local Institution - 0325, Sofia
- Canada (3):
  - Local Institution - 0002, Halifax, Nova Scotia
  - Local Institution - 0178, Ottawa, Ontario
  - Local Institution - 0156, Toronto, Ontario
- Chile (6):
  - Local Institution - 0361, Antofagasta, AN
  - Local Institution - 0302, Las Condes, Arica y Parinacota Region
  - Local Institution - 0222, Santiago, Santiago Metropolitan
  - Local Institution - 0199, Santiago, Santiago Metropolitan
  - Local Institution - 0293, Concepción
  - Local Institution - 0150, Independencia
- China (24):
  - Local Institution - 0175, Beijing, Beijing Municipality
  - Local Institution - 0167, Fuzhou, Fujian
  - Local Institution - 0141, Xiamen, Fujian
  - Local Institution - 0327, Zhangzhou, Fujian
  - Local Institution - 0312, Guangzhou, Guangdong
  - Local Institution - 0210, Shantou, Guangdong
  - Local Institution - 0255, Nanning, Guangxi
  - Local Institution - 0317, Harbin, Heilongjiang
  - Local Institution - 0004, Changsha, Hunan
  - Local Institution - 0117, Nanjing, Jiangsu
  - Local Institution - 0316, Nanjing, Jiangsu
  - Local Institution - 0023, Nanchang, Jiangxi
  - Local Institution - 0177, Shenyang, Liaoning
  - Local Institution - 0014, Xi'an, Shaanxi
  - Local Institution - 0359, Jinan, Shandong
  - Local Institution - 0123, Linyi, Shandong
  - Local Institution - 0185, Shanghai, Shanghai Municipality
  - Local Institution - 0212, Shanghai Shi, Shanghai Municipality
  - Local Institution - 0246, Chengdu, Sichuan
  - Local Institution - 0183, Hangzhou, Zhejiang
  - Local Institution - 0089, Hangzhou, Zhejiang
  - Local Institution - 0113, Beijing
  - Local Institution - 0122, Shanghai Shi
  - Local Institution - 0046, Zhengzhou
- Colombia (4):
  - Local Institution - 0310, Rionegro, Antioquia
  - Local Institution - 0328, Barranquilla, Atlántico
  - Local Institution - 0218, Bogotá
  - Local Institution - 0307, Medellín
- Czechia (4):
  - Local Institution - 0092, Ostrava, Moravian-Silesian
  - Local Institution - 0129, Pilsen, Plzeň Region
  - Local Institution - 0243, Hradec Králové
  - Local Institution - 0236, Olomouc
- Finland (3):
  - Local Institution - 0060, Kuopio, Northern Savonia
  - Local Institution - 0171, Tampere
  - Local Institution - 0126, Vaasa
- France (12):
  - Local Institution - 0162, Lille, Hauts-de-France
  - Local Institution - 0144, La Tronche, Isère
  - Local Institution - 0059, Toulouse, Midi-Pyrénées
  - Local Institution - 0390, Brest
  - Local Institution - 0054, Limoges
  - Local Institution - 0151, Marseille
  - Local Institution - 0239, Montpellier
  - Local Institution - 0206, Paris
  - Local Institution - 0207, Paris
  - Local Institution - 0130, Pessac
  - Local Institution - 0400, Reims
  - Local Institution - 0057, Saint-Herblain
- Germany (14):
  - Local Institution - 0072, Wangen, Baden-Wurttemberg
  - Local Institution - 0270, Landshut, Bavaria
  - Local Institution - 0024, Rosenheim, Bavaria
  - Local Institution - 0187, Solingen, North Rhine-Westphalia
  - Local Institution - 0172, Kiel, Schleswig-Holstein
  - Local Institution - 0231, Berlin
  - Local Institution - 0158, Braunschweig
  - Local Institution - 0157, Erfurt
  - Local Institution - 0073, Essen
  - Local Institution - 0103, Gera
  - Local Institution - 0071, Göttingen
  - Local Institution - 0357, Kaiserslautern
  - Local Institution - 0264, Münster
  - Local Institution - 0083, Sindelfingen
- Hungary (5):
  - Local Institution - 0240, Budapest
  - Local Institution - 0234, Budapest
  - Local Institution - 0012, Farkasgyepű
  - Local Institution - 0244, Mátraháza
  - Local Institution - 0241, Szolnok
- India (7):
  - Local Institution - 0303, Eluru, Andhra Pradesh
  - Local Institution - 0319, Visakhapatnam, Andhra Pradesh
  - Local Institution - 0008, Nagpur, Maharashtra
  - Local Institution - 0125, Dwarka, National Capital Territory of Delhi
  - Local Institution - 0020, Hyderabad, Telangana
  - Local Institution - 0078, Delhi
  - Local Institution - 0036, Pune
- Italy (8):
  - Local Institution - 0281, Ferrara (Cona), Emilia-Romagna
  - Local Institution - 0174, Novara, Piedmont
  - Local Institution - 0279, Catania, Sicily
  - Local Institution - 0194, Aviano (PN)
  - Local Institution - 0032, Candiolo
  - Local Institution - 0111, Genova
  - Local Institution - 0033, Milan
  - Local Institution - 0040, Napoli
- Japan (17):
  - Local Institution - 0055, Toyohashi, Aichi-ken
  - Local Institution - 0363, Aomori, Aomori
  - Local Institution - 0258, Funabashi, Chiba
  - Local Institution - 0256, Tōon, Ehime
  - Local Institution - 0251, Nishinomiya-shi, Hyōgo
  - Local Institution - 0056, Kanazawa, Ishikawa-ken
  - Local Institution - 0259, Kamakura, Kanagawa
  - Local Institution - 0248, Kumamoto, Kumamoto
  - Local Institution - 0254, Sendai, Miyagi
  - Local Institution - 0250, Osakasayama-shi, Osaka
  - Local Institution - 0247, Koshigaya, Saitama
  - Local Institution - 0166, Hidaka, Saitama-Pref
  - Local Institution - 0253, Hamamatsu
  - Local Institution - 0252, Hirakata-shi
  - Local Institution - 0341, Hiroshima
  - Local Institution - 0257, Sendai
  - Local Institution - 0249, Yokohama
- Malaysia (3):
  - Local Institution - 0275, George Town, Pulau Pinang
  - Local Institution - 0271, Kuching, Sarawak
  - Local Institution - 0277, Kuala Lumpur
- Mexico (6):
  - Local Institution - 0070, Zapopan, Jalisco
  - Local Institution - 0075, Mexico City, Mexico City
  - Local Institution - 0386, Monterrey, Nuevo León
  - Local Institution - 0385, Mexico City
  - Local Institution - 0097, Oaxaca City
  - Local Institution - 0124, Querétaro
- Netherlands (6):
  - Local Institution - 0286, Breda, North Brabant
  - Local Institution - 0100, 's-Hertogenbosch
  - Local Institution - 0161, Amersfoort
  - Local Institution - 0261, Deventer
  - Local Institution - 0110, Nijmegen
  - Local Institution - 0094, Tilburg
- Norway (2):
  - Local Institution - 0164, Grålum, Akershus
  - Local Institution - 0050, Drammen, Buskerud
- Peru (3):
  - Local Institution - 0121, San Borja, Lima region
  - Local Institution - 0155, Lima
  - Local Institution - 0296, Lima
- Poland (5):
  - Local Institution - 0227, Przemyśl, Podkarpackie Voivodeship
  - Local Institution - 0329, Katowice
  - Local Institution - 0186, Lodz
  - Local Institution - 0041, Opole
  - Local Institution - 0105, Warsaw
- Portugal (2):
  - Local Institution - 0294, Braga
  - Local Institution - 0278, Lisbon
- Romania (9):
  - Local Institution - 0191, Baloteşti, Ilfov
  - Local Institution - 0044, Bucharest
  - Local Institution - 0049, Bucharest
  - Local Institution - 0136, Bucharest
  - Local Institution - 0209, Cluj-Napoca
  - Local Institution - 0084, Craiova
  - Local Institution - 0132, Floresti/ Cluj
  - Local Institution - 0127, Iași
  - Local Institution - 0068, Iași
- Singapore (2):
  - Local Institution - 0267, Singapore
  - Local Institution - 0269, Singapore
- South Korea (4):
  - Local Institution - 0343, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0336, Deagu, Taegu-Kwangyǒkshi
  - Local Institution - 0335, Junggu, Taejǒn-Kwangyǒkshi
  - Local Institution - 0342, Yangsan
- Spain (9):
  - Local Institution - 0181, Málaga, Málaga
  - Local Institution - 0074, Barakaldo
  - Local Institution - 0009, Barcelona
  - Local Institution - 0142, Barcelona
  - Local Institution - 0099, Jaén
  - Local Institution - 0266, Madrid
  - Local Institution - 0021, Madrid
  - Local Institution - 0179, Madrid
  - Local Institution - 0263, Murcia
- Sweden (2):
  - Local Institution - 0039, Stockholm, Stockholm County
  - Local Institution - 0010, Gävle
- Switzerland (4):
  - Local Institution - 0399, Lausanne
  - Local Institution - 0053, Sankt Gallen
  - Local Institution - 0019, Thun
  - Local Institution - 0262, Villars-sur-Glâne
- Taiwan (5):
  - Local Institution - 0389, Kaohsuing City, Kaohsiung
  - Local Institution - 0388, Taoyuan, Taoyuan
  - Local Institution - 0203, Chiayi City
  - Local Institution - 0387, Kaohsiung City
  - Local Institution - 0035, New Taipei City
- Thailand (3):
  - Local Institution - 0272, Bangkok
  - Local Institution - 0273, Khon Kaen
  - Local Institution - 0274, Songkhla
- Turkey (Türkiye) (10):
  - Local Institution - 0107, Istanbul, Bagcilar
  - Local Institution - 0242, Adana
  - Local Institution - 0091, Adana
  - Local Institution - 0118, Antalya
  - Local Institution - 0238, Çankaya
  - Local Institution - 0017, Istanbul
  - Local Institution - 0133, Istanbul
  - Local Institution - 0367, Istanbul
  - Local Institution - 0364, Izmir
  - Local Institution - 0235, Karşıyaka
- United Kingdom (7):
  - Local Institution - 0365, Aberdeen, Aberdeenshire
  - Local Institution - 0112, Middlesbrough, Cleveland
  - Local Institution - 0114, Cambridge
  - Local Institution - 0182, Cardiff
  - Local Institution - 0007, Guildford
  - Local Institution - 0087, London
  - Local Institution - 0371, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07361510.html